CLINICAL TRIAL: NCT00124150
Title: Phase 3 Study (Multi-center, Randomized Controlled Clinical Trial) of Intravenous Magnesium Sulfate to Improve Outcome After Aneurysmal Subarachnoid Haemorrhage
Brief Title: Intravenous Magnesium Sulfate in Aneurysmal Subarachnoid Haemorrhage (IMASH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: George KC WONG, Division of Neurosurgery, The Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IMASH trial
Record Dates: First submitted 2005-07-26; First posted 2005-07-27 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-07

CONDITIONS: Subarachnoid Hemorrhage
Keywords: subarachnoid hemorrhage; magnesium sulfate
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- M (Experimental): Intravenous magnesium sulfate infusion for 14 days.
  Interventions: Drug: Intravenous magnesium sulfate infusion
- S (No Intervention): Saline infusion without additional magnesium sulfate.

INTERVENTIONS:
Drug: Intravenous magnesium sulfate infusion — 80mg per day
  Arms: M

SUMMARY:
The IMASH trial is a simple, randomized, double-blinded, placebo-controlled, multi-center trial to answer the question: "Does intravenous magnesium sulfate improve clinical outcome after aneurysmal subarachnoid hemorrhage?"

DETAILED DESCRIPTION:
Vasospasm worsen outcome in patients with aneurysmal subarachnoid hemorrhage (ASAH).

Magnesium is known to dilate cerebral arteries and to block N-methyl-D-aspartate receptors in the injured neurons.

Intravenous magnesium may prevent vasospasm after subarachnoid hemorrhage and may protect neurons against damage during established vasospasm.

The IMASH trial is a randomized, placebo-controlled, double-blinded, multi-center trial to evaluate the effect that intravenous magnesium sulfate infusion on the clinical outcome of patients with aneurysmal subarachnoid haemorrhage.

Methods:

After obtaining randomisation code:

* Start MgSO4 20 mmol over 30 minutes, followed by infusion of 80 mmol/day or equivalent volume of saline within 48 h after onset of symptom,
* Study drug to be infused for 14 days from the day of hemorrhage (regarded as day 0).
* Measure plasma magnesium concentration daily and perform transcranial Doppler to monitor blood flow velocities of both middle cerebral arteries and extracranial segment of the internal carotid arteries.
* Plasma magnesium concentration in the IV MgSO4 group should be raised to 2.0-2.5 mmol/L or twice the serum baseline level. Patients that are randomized to saline infusion will only have their magnesium levels normalized if there is a clinical indication to do so.

Outcome assessment Primary outcome: Extended Glasgow Outcome Scale at six months Secondary outcome: Incidence of clinical vasospasm, Barthel Index; modified Rankin score, modified National Institute of Health Stroke Score, MCA velocities, other major complications

Study duration:

6 years with a refined sample size of 340 after analysis of pilot study data; with planned interim analysis.

ELIGIBILITY:
Inclusion Criteria:

* ASAH (as indicated by CT scan or lumbar puncture and an intracranial aneurysm confirmed by computer tomographic or conventional angiography)
* Within 48 hrs of ictus (hemorrhage event)

Exclusion Criteria:

* Pregnancy
* Major renal, hepatic or pulmonary disease
* Major cardiac disease or recent myocardial infarct (< 6 months)
* Age less than 18 years
* Moribund condition on admission (defined as a patient that is in such a poor clinical condition that further active neurosurgical management would not be anticipated)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2002-06; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Extended Glasgow Outcome Scale | At six months

SECONDARY OUTCOMES:
Incidence of clinical vasospasm | Within first 14 days
Barthel Index | At six months
Modified Rankin Score | At six months
Modified National Institute of Health Stroke Score | At six months
Other major complications requiring intensive care unit admission | During first 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Wai S Poon, MB ChB FRCS, Principal Investigator — Department of Surgery, The Chinese University of Hong Kong
Locations (1):
- Department of Surgery, The Chinese University of Hong Kong, Hong Kong, China

REFERENCES:
- [Background] Boet R, Mee E. Magnesium sulfate in the management of patients with Fisher Grade 3 subarachnoid hemorrhage: a pilot study. Neurosurgery. 2000 Sep;47(3):602-6; discussion 606-7. doi: 10.1097/00006123-200009000-00014. PMID 10981747
- [Background] Boet R, Poon WS, Chan MT. Re: Magnesium: a useful adjunct in the prevention of cerebral vasospasm following aneurysmal subarachnoid haemorrhage. J Clin Neurosci. 2003 May;10(3):394. doi: 10.1016/s0967-5868(03)00006-7. No abstract available. PMID 12763359
- [Background] Wong GK, Poon WS, Chan MT, Boet R, Gin T, Lam CW. The effect of intravenous magnesium sulfate infusion on serum levels of sodium and potassium in patients with aneurysmal subarachnoid hemorrhage. Magnes Res. 2007 Mar;20(1):37-42. PMID 17536487
- [Result] Boet R, Chan MT, Poon WS, Wong GK, Wong HT, Gin T. Intravenous magnesium sulfate to improve outcome after aneurysmal subarachnoid hemorrhage: interim report from a pilot study. Acta Neurochir Suppl. 2005;95:263-4. doi: 10.1007/3-211-32318-x_53. PMID 16463861
- [Result] Wong GK, Chan MT, Boet R, Poon WS, Gin T. Intravenous magnesium sulfate after aneurysmal subarachnoid hemorrhage: a prospective randomized pilot study. J Neurosurg Anesthesiol. 2006 Apr;18(2):142-8. doi: 10.1097/00008506-200604000-00009. PMID 16628069
- [Result] Wong GK, Chan MT, Poon WS, Boet R, Gin T. Magnesium therapy within 48 hours of an aneurysmal subarachnoid hemorrhage: neuro-panacea. Neurol Res. 2006 Jun;28(4):431-5. doi: 10.1179/016164106X115035. PMID 16759446
- [Result] Wong GK, Chan MT, Boet R, Poon WS. Correspondence to 'dose evaluation for long-term magnesium treatment in aneurysmal subarachnoid haemorrhage'. J Clin Pharm Ther. 2006 Aug;31(4):407. doi: 10.1111/j.1365-2710.2006.00728.x. No abstract available. PMID 16882114
- [Derived] Wong GK, Poon WS. Clinical, transcranial Doppler ultrasound, radiological features and, prognostic significance of delayed cerebral ischemia. Acta Neurochir Suppl. 2013;115:9-11. doi: 10.1007/978-3-7091-1192-5_3. PMID 22890635
- [Derived] Wong GK, Poon WS, Boet R, Chan MT, Gin T, Ng SC, Zee BC. Health-related quality of life after aneurysmal subarachnoid hemorrhage: profile and clinical factors. Neurosurgery. 2011 Jun;68(6):1556-61; discussion 1561. doi: 10.1227/NEU.0b013e31820cd40d. PMID 21311383
- [Derived] Wong GK, Poon WS, Chan MT, Boet R, Gin T, Ng SC, Zee BC; IMASH Investigators. Intravenous magnesium sulphate for aneurysmal subarachnoid hemorrhage (IMASH): a randomized, double-blinded, placebo-controlled, multicenter phase III trial. Stroke. 2010 May;41(5):921-6. doi: 10.1161/STROKEAHA.109.571125. Epub 2010 Apr 8. PMID 20378868